CLINICAL TRIAL: NCT05034926
Title: A Multinational, Non-Interventional, Prospective Study of Nivolumab (BMS-936558) in Patients With Locally Advanced or Metastatic (Stage IIIB-IV) Non-Small Cell Lung Cancer (NSCLC) With Squamous and Non-Squamous Histology After Prior Chemotherapy Treated in Real World Settings in Greece and Cyprus - The 'Lucence' Study
Brief Title: A Study of Nivolumab in Participants With Locally Advanced or Metastatic (Stage IIIB-IV) Non-Small Cell Lung Cancer (NSCLC) With Squamous and Non-Squamous Histology After Prior Chemotherapy Treated in Real World Settings in Greece and Cyprus
Acronym: LUCENCE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7U9
Record Dates: First submitted 2021-08-16; First posted 2021-09-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: BMS-936558; Greece; Cyprus; Locally advanced; Metastatic NSCLC; Nivolumab; OPDIVO®; Prospective Study; Stage IIIb/IV; 2nd line treatment; 3rd line treatment; Observational study; LUCENCE study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with locally advanced or metastatic (stage IIIB-IV) non-small cell lung cancer (NSCLC)

SUMMARY:
The purpose of this observational study is to estimate the overall survival (OS) rates in the overall study population treated with nivolumab in the second and third line setting in real world clinical practice in Greece and Cyprus. The study is descriptive in nature and is not planned to reject or affirm any formal statistical hypothesis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female adult Greek-speaking patients, of any race (residing in Greece or Cyprus), aged at least 18 years at time of initiation of nivolumab treatment.
* Histologically- or cytologically-confirmed diagnosis of locally advanced or metastatic (stage IIIB-IV) Non-Small Cell Lung Cancer (NSCLC) with Squamous Cell Carcinoma (SCC) or Non-Squamous Cell Carcinoma (NSCC) histological subtype
* Initiated on second or third line treatment with nivolumab as monotherapy after prior chemotherapy as per the product's Summary of Product Characteristics (SmPC) prior to informed consent obtainment, and for whom therapy is ongoing and no more than one infusion has been administered from treatment initiation to obtaining the signed informed consent
* Decision to prescribe nivolumab treatment has been taken prior to their enrollment in the study and is clearly separated from the physician's decision to include the patient in the current study
* Provided signed informed consent for participating in the study and for collecting and analyzing medical data pertinent to the objectives of this study

Exclusion Criteria:

* Current primary diagnosis of a cancer other than NSCLC that requires systemic or other treatment
* Previously treated with nivolumab or other non-chemotherapy agents, with the exception of immune checkpoint inhibitors (anti-PD-1(Programmed cell death-1)/anti-PD-L1 (Programmed death-ligand 1) agent, other than nivolumab) administered in combination with chemotherapy
* Currently receiving or are planned to receive treatment with any investigational drug/device/intervention or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to nivolumab therapy initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 350 locally advanced/metastatic NSCLC patients who are eligible for participation in the study according to the inclusion and exclusion criteria are planned to be enrolled over a 24-month recruitment period by approximately 27 lung cancer specialists practicing in the public or private healthcare sector throughout Greece and Cyprus.
  Patients treated with nivolumab in the second and third line setting in real world clinical practice and who are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants surviving at the landmark timepoint of 12 months after the initiation of nivolumab treatment, in the overall study population | Up to 12 months
Proportion of participants surviving at the landmark timepoint of 24 months after the initiation of nivolumab treatment, in the overall study population | Up to 24 months
Proportion of participants surviving at the landmark timepoint of 36 months after the initiation of nivolumab treatment, in the overall study population | Up to 36 months

SECONDARY OUTCOMES:
Proportion of participants surviving at the landmark timepoint 12 months after the initiation of nivolumab treatment, among the Squamous Cell Carcinoma (SCC) subpopulation | Up to 12 months
Proportion of participants surviving at the landmark timepoint 24 months after the initiation of nivolumab treatment, among the SCC subpopulation | Up to 24 months
Proportion of participants surviving at the landmark timepoint 36 months after the initiation of nivolumab treatment, among the SCC subpopulation | Up to 36 months
Proportion of participants surviving at the landmark timepoint 12 months after the initiation of nivolumab treatment, among the Non-Squamous Cell Carcinoma (NSCC) subpopulation | Up to 12 months
Proportion of participants surviving at the landmark timepoint 24 months after the initiation of nivolumab treatment, among the NSCC subpopulation | Up to 24 months
Proportion of participants surviving at the landmark timepoint 36 months after the initiation of nivolumab treatment, among the NSCC subpopulation | Up to 36 months
Proportion of participants surviving at the landmark timepoint 12 months after the initiation of nivolumab treatment per line of nivolumab treatment | Up to 12 months
Proportion of participants surviving at the landmark timepoint 24 months after the initiation of nivolumab treatment per line of nivolumab treatment | Up to 24 months
Proportion of participants surviving at the landmark timepoint 36 months after the initiation of nivolumab treatment per line of nivolumab treatment | Up to 36 months
Proportion of participants who have not progressed or died from any cause at the landmark timepoint 12 months after the initiation of nivolumab treatment | Up to 12 months
Proportion of participants who have not progressed or died from any cause at the landmark timepoint 24 months after the initiation of nivolumab treatment | Up to 24 months
Proportion of participants who have not progressed or died from any cause at the landmark timepoint 36 months after the initiation of nivolumab treatment | Up to 36 months
Proportion of participants with an investigator-assessed best overall response (BOR) of either a confirmed complete response (CR) or confirmed PR (ORR rate) at the landmark timepoint of 12 months after the initiation of nivolumab treatment | Up to 12 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Proportion of participants with an investigator-assessed BOR of confirmed CR or PR or stable disease (SD) (DCR rate), at the landmark timepoint of 12 months after the initiation of nivolumab treatment | Up to 12 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Time from start of nivolumab treatment to the first documented investigator-assessed response (CR or PR) (i.e., TTR), among participants who achieved at least PR | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Time from start of nivolumab treatment to best response (e.g., if a participant had both PR and CR, time to CR), among participants who achieved at least PR | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab.
Kaplan-Meier estimated median time from first documented response (CR or PR) to the date of first documented progression or death (due to any cause in the absence of progression), among participants who achieved at least PR (i.e., DoR) | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab.
Kaplan-Meier estimated median time from best response (e.g., if a patient had both PR and CR, time from CR) to the date of first documented progression or death (due to any cause in the absence of progression), among patients who achieved at least PR | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab.
Frequencies of baseline participant and disease characteristics of interest | Up to approximately 59 months
  This refers to the overall study population and the SCC and NSCC subpopulation.
Distribution of associations of baseline participant and disease characteristics with survival at 36 months post-treatment initiation | Up to 36 months
Distribution of the number of nivolumab doses administered | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Distribution of the rate of dose modifications (including dose delays/withholdings) | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Distribution of the rate of permanent treatment discontinuation | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Distribution of the frequencies of reasons for dose modifications/discontinuations | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Distribution of the types and frequencies of next treatment planned to be administered for NSCLC after nivolumab discontinuation | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Kaplan-Meier estimated time from nivolumab treatment initiation until discontinuation due to any reason | Up to approximately 59 months
  This refers to the overall study population, the SCC and NSCC subpopulations, and the subpopulations per line of nivolumab treatment.
Distribution of exposure-adjusted incidence rate (EAIR), severity (grade), and management of the specified types of treatment-related AEs in the overall study population | Up to approximately 59 months
Time to onset of high-grade (Grade 3 or higher) immune-related adverse events (irAEs) per AE category | Up to approximately 59 months
Time to resolution of high-grade (Grade 3 or higher) irAEs per AE category | Up to approximately 59 months
Incidence of adverse events leading to nivolumab treatment permanent discontinuation, in the overall study population | Up to approximately 59 months
Distribution of type of adverse events leading to nivolumab treatment permanent discontinuation, in the overall study population | Up to approximately 59 months
Change in the total LCSS score in the overall study population | Up to approximately 59 months
Change in the total ASBI score throughout the study observation period examined using longitudinal analysis | Up to approximately 59 months
Change in the total Average Symptom Burden Index (ASBI) score, in the overall study population | Up to approximately 59 months
  In addition, change in the total ASBI score throughout the study observation period will be examined using longitudinal analysis
Change in the individual domain scores from baseline to each post-baseline predefined timepoint in the overall study population | Up to approximately 59 months
Symptom improvement rate, at the post-baseline predefined timepoints, using the Lung Cancer Symptom Scale (LCSS) Average Symptom Burden Index (ASBI), in the overall study population | Up to approximately 59 months
Change in the EuroQol (EQ-5D) utility index score, from baseline at the post-baseline predefined timepoints, in the overall study population | Up to approximately 59 months
Change in the EuroQol Visual Analogue Scale (EQ-VAS) score, from baseline at the post-baseline predefined timepoints, in the overall study population | Up to approximately 59 months
Change in the proportion of participants in the five-level version of the EuroQol five-dimensional questionnaire (EQ-5D-5L) dimension levels (no problems, with problems) from baseline at the post-baseline predefined timepoints | Up to approximately 59 months
  in the overall study population
Distribution of Person-time incidence rate (per 100 participant-weeks) of inpatient hospitalizations for the management of treatment-related AEs, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Emergency room attendances for the management of treatment-related AEs, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Hospital outpatient visits for the management of treatment-related AEs, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Visits at office-based physicians for the management of treatment-related AEs, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Home visits by physicians, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Length of hospital stay, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Types and frequencies of medical procedures/interventions/diagnostic testing utilization, during the entire study observation period, in the overall study population | Up to approximately 59 months
Distribution of Prescribed medications for the management of treatment-related AEs, during the entire study observation period, in the overall study population | Up to approximately 59 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution - 0002, Stróvolos, Cyprus
- Local Institution - 0001, Athens, Greece

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm